CLINICAL TRIAL: NCT01183715
Title: A Phase 1 Placebo-Controlled Study To Assess The Safety, Tolerability And Pharmacokinetics Of PF-05161704 After Administration Of Single Escalating Oral Doses Under Fed And Fasted Conditions In Healthy Volunteers
Brief Title: A Single Dose Study Of PF-05161704 In Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: B2911001
Record Dates: First submitted 2010-08-13; First posted 2010-08-18 (Estimated); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Single Ascending Dose; Phase 1; Safety and Tolerability; PK; Healthy Subjects
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort 1 (Experimental): Subjects in Cohort 1 will receive 2 single doses of PF-05161704 and 1 placebo dose in random order in Periods 1-3; in addition, 1 dose of PF-05161704 will be administered in Period 4 in the fasted state.
  Interventions: Drug: PF-05161704 or placebo
- Cohort 2 (Experimental): Subjects in Cohort 2 will receive 2 single doses of PF-05161704 and 1 placebo dose in random order in Periods 1-3
  Interventions: Drug: PF-05161704 or placebo

INTERVENTIONS:
Drug: PF-05161704 or placebo — PF-05161704 will be administered as an extemporaneously prepared suspension in the initially planned dose range of 1.5 mg to 300 mg. Correspondingly, placebo doses will be administered as suspension
  Arms: Cohort 1
Drug: PF-05161704 or placebo — PF-05161704 will be administered as an extemporaneously prepared suspension in the initially planned dose range of 1.5 mg to 300 mg. Correspondingly, placebo doses will be administered as suspension
  Arms: Cohort 2

SUMMARY:
The primary purpose of this study is to evaluate the safety, tolerability and pharmacokinetics of single oral doses of PF-05161704 in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female (non child-bearing potential) subjects between the ages of 18 and 55 years, inclusive (Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12-lead ECG and clinical laboratory tests).
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lbs).

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* Any condition possibly affecting drug absorption (eg, gastrectomy).
* History of regular alcohol consumption exceeding 7 drinks/week for females or 14 drinks/week for males (1 drink = 5 ounces (150 mL) of wine or 12 ounces (360 mL) of beer or 1.5 ounces (45 mL) of hard liquor) within 6 months of screening.
* History or evidence of habitual use of tobacco or nicotine containing products within 3 months of Screening or positive cotinine test at screening or Day 0 of period one

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2010-07; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of escalating single oral doses of PF-05161704 in healthy subjects | 1 month
Single dose pharmacokinetics of PF-05161704 and its metabolite PF-05200145 | 1 month

SECONDARY OUTCOMES:
Preliminary pharmacodynamics of PF-05161704 | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B2911001&StudyName=A%20Single%20Dose%20Study%20Of%20PF-05161704%20In%20Healthy%20Volunteers